CLINICAL TRIAL: NCT06099522
Title: Internet-based Cognitive Behavioral Treatment for Gambling Disorder - a Randomized Controlled Trial
Brief Title: Internet-CBT for Gambling Disorder - a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Deakin University (Other)
Responsible Party: Principal Investigator, Olof Molander, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2023-01075-01
Record Dates: First submitted 2023-08-29; First posted 2023-10-25 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either standard iCBT and "Spelpaus" (treatment condition), or "Spelpaus" only (control condition).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based cognitive behavioral therapy (iCBT) (Experimental): An 8-module internet-delivered cognitive behavioral therapy program. Participants receiving treatment will simultaneously use "Spelpaus" - a self-exclusion gambling service.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy (iCBT)
- "Spelpaus" (gambling self-exclusion) (No Intervention): "Spelpaus" only - a self-exclusion gambling service.

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy (iCBT) — The treatment is a newly developed iCBT 8 module program, with interventions targeting gambling-related loss of control, through 4 clinical processes: Gambling triggers, Gambling-related anticipation, the Gambling zone and Chasing behaviors. The treatment will be delivered with therapist support.
  Arms: Internet-based cognitive behavioral therapy (iCBT)

SUMMARY:
The study is a randomized controlled trial (Total N=150; each condition n=75) of internet-based cognitive behavioral therapy (iCBT), with measures at pre, weekly during treatment, post, three and at six month follow-up. Participants will be assigned to either standard iCBT and "Spelpaus" (treatment condition), or "Spelpaus" only (control condition).

DETAILED DESCRIPTION:
Recruitment will be done through online advertisement via social media and gambling-related websites. Participants will self-referred to the study via a study dedicated website (www.spelstudien.se). Login to a treatment platform will be verified using double authentication (detailed description of the online platform is provided in the application to the Swedish Ethical Review Authority). Written information about the study will be provided on the web page. Consent will be done online, with the possibility for participants to download study information and consent. Consenting participants will start a screening procedure. After screening, participants will be contacted for a telephone assessment with a clinical psychologist. During this interview, participants will be assessed for GD with a diagnostic interview, as well as the inclusion criteria for utilization of "Spelpaus". If meeting criteria for the study, participants will be referred to the baseline/pre-measures - which will start with an additional informed consent for the treatment phase and the iCBT. Inclusion will be done after the completion of the informed consent and baseline/pre-measures. After that, participant will be randomized to iCBT and "Spelpaus" (treatment condition), or "Spelpaus" only (control condition). Randomization will be conducted by a third party using a true random service, https://random.org. Participants assigned to the control condition in the randomized controlled trial will receive a voucher of total 1000 Swedish Krona's when completing the post and follow up measures. Participants assigned to the control condition in the randomized controlled trial will receive a voucher of total 1000 Swedish Krona's when completing the post and follow up measures.

ELIGIBILITY:
Inclusion Criteria:

* Screen positive for GD, as measured with the Gambling Disorder Identification Test (total score ≥20 GDIT).
* Fulfilling GD, assessed according to the Structured Clinical Interview for Gambling Disorder (SCI-GD).
* Utilization of "Spelpaus", 3 months from treatment start.
* ≥18 years of age.
* Able to provide digital informed consent.

Exclusion Criteria:

* Other ongoing psychological treatment for GD.
* Severe depression, screened according to the Montgomery Åsberg Depression Rating Scale (total score >34 MADRS-S).
* Suicidality, screening of ≥4 points on item 9 of the MADRS-S

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The Gambling Symptom Assessment Scale | 6 month after treatment cessation
  Primary outcome will be gambling symptoms, measured with the the Gambling Symptom Assessment Scale. Minimum score is 0 and maximum score is 48, with higher scores indicated higher frequency of gambling symptoms.

SECONDARY OUTCOMES:
The TimeLine Followback for gambling | 6 month after treatment cessation
  Gambling behavior (days per week gambled) will be measured with a self-report item adapted from the TimeLine Followback for gambling.
The Generalized Anxiety Disorder 7-itemscale | 6 month after treatment cessation
  Anxiety symptoms will be measured by the Generalized Anxiety Disorder 7-itemscale.
The Patient Health Questionnaire | 6 month after treatment cessation
  Depressive symptoms will be measured with the The Patient Health Questionnaire.
The Alcohol Use Disorders Identification Test | 6 month after treatment cessation
  Alcohol problems will be measured with the Alcohol Use Disorders Identification Test.
The Drug Use Disorders Identification Test | 6 month after treatment cessation
  Drug problems will be measured with the Drug Use Disorders Identification Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for psychiatry research, Stockholm, Sweden